CLINICAL TRIAL: NCT02011126
Title: A Phase II Study of Imetelstat (GRN163L, NSC# 754228) in Children With Relapsed or Refractory Solid Tumors
Brief Title: Imetelstat Sodium in Treating Younger Patients With Relapsed or Refractory Solid Tumors
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: IND no longer available.
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADVL1321; NCI-2013-01640 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ADVL1321 (Other: Childrens Oncology Group); ADVL1321 (Other: CTEP); U10CA098543 (NIH)
Record Dates: First submitted 2013-12-10; First posted 2013-12-13 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2014-05

CONDITIONS: Hepatoblastoma; Previously Treated Childhood Rhabdomyosarcoma; Recurrent Childhood Liver Cancer; Recurrent Childhood Rhabdomyosarcoma; Recurrent Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor; Recurrent Neuroblastoma; Recurrent Osteosarcoma; Rhabdomyosarcoma
MeSH Terms: conditions — Hepatoblastoma; Neuroectodermal Tumors, Primitive, Peripheral; Neuroblastoma; Osteosarcoma; Rhabdomyosarcoma | interventions — imetelstat; GRN163L peptide

ARMS (1):
- Treatment (imetelstat sodium) (Experimental): Patients receive imetelstat sodium IV over 2 hours on days 1 and 8. Treatment repeats every 21 days for up to 36 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Imetelstat Sodium; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Imetelstat Sodium — Given IV
  Other Names: GRN163L; GRN163L, Sodium Salt
Other: Laboratory Biomarker Analysis — Optional correlative studies

SUMMARY:
This phase II trial studies the side effects and how well imetelstat sodium works in treating younger patients with relapsed or refractory solid tumors. Imetelstat sodium may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the objective response rate, defined as partial response or better, of imetelstat (imetelstat sodium) in children with relapsed or refractory solid tumors.

II. To further define and describe the toxicities associated with imetelstat in children with recurrent/refractory solid tumors.

SECONDARY OBJECTIVES:

I. To determine the time to progression following treatment with imetelstat in children with relapsed or refractory solid tumors.

TERTIARY OBJECTIVES:

I. To measure tumor telomere length in archival samples, and to correlate telomere length to the clinical outcome of the study.

OUTLINE:

Patients receive imetelstat sodium intravenously (IV) over 2 hours on days 1 and 8. Treatment repeats every 21 days for up to 36 courses in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with any of the following tumors who have relapsed or refractory disease are eligible:

  * Osteosarcoma
  * Ewing?s sarcoma / peripheral primitive neuroectodermal tumor (PNET)
  * Rhabdomyosarcoma
  * Neuroblastoma (measurable or evaluable disease)
  * Hepatoblastoma
* Patients must have had histologic verification of malignancy at original diagnosis or relapse
* Patients must have radiographically measurable disease (with the exception of neuroblastoma)

  * Measurable disease is defined as the presence of at least one lesion on magnetic resonance imaging (MRI) or computed tomography (CT) scan that can be accurately measured with the longest diameter a minimum of 10 mm in at least one dimension (CT scan slice thickness no greater than 5 mm)
  * Note: the following do not qualify as measurable disease:

    * Malignant fluid collections (e.g., ascites, pleural effusions)
    * Bone marrow infiltration
    * Lesions only detected by nuclear medicine studies (e.g., bone, gallium or positron emission tomography [PET] scans) except as defined below for neuroblastoma
    * Elevated tumor markers in plasma or cerebrospinal fluid (CSF)
    * Previously radiated lesions that have not demonstrated clear progression post radiation
    * Leptomeningeal lesions that do not meet the measurements noted above
* Patients with neuroblastoma who do not have measurable disease but have evaluable disease on 131I-metaiodobenzylguanidine (MIBG) scans are eligible
* Patients must have a Lansky or Karnofsky performance status score of >= 50, corresponding to Eastern Cooperative Oncology Group (ECOG) categories 0, 1 or 2; use Karnofsky for patients > 16 years of age and Lansky for patients =< 16 years of age; patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study
* Myelosuppressive chemotherapy: patients with solid tumors must not have received myelosuppressive chemotherapy within 3 weeks of enrollment onto this study (6 weeks if prior nitrosourea)
* Hematopoietic growth factors: at least 7 days must have elapsed since the completion of therapy with a growth factor; at least 14 days must have elapsed after receiving pegfilgrastim
* Biologic (anti-neoplastic agent): at least 7 days must have elapsed since completion of therapy with a biologic agent; for agents that have known adverse events occurring beyond 7 days after administration, this period prior to enrollment must be extended beyond the time during which adverse events are known to occur
* Monoclonal antibodies: at least 3 half-lives must have elapsed since prior therapy that included a monoclonal antibody
* Radiotherapy: >= 2 weeks must have elapsed since local palliative radiation therapy (XRT) (small port); >= 6 weeks must have elapsed since treatment with therapeutic doses of MIBG; >= 3 months must have elapsed if prior craniospinal XRT was received, if >= 50% of the pelvis was irradiated, or if total body irradiation (TBI) was received; >= 6 weeks must have elapsed if other substantial bone marrow irradiation was given
* Stem cell transplant or rescue without TBI: no evidence of active graft versus (vs.) host disease and >= 2 months must have elapsed since transplant
* For patients with solid tumors without bone marrow involvement:

  * Peripheral absolute neutrophil count (ANC) >= 1000/uL
* For patients with solid tumors without bone marrow involvement:

  * Platelet count >= 100,000/uL (transfusion independent, defined as not receiving platelet transfusions within a 7 day period prior to enrollment)
* For patients with solid tumors without bone marrow involvement:

  * Hemoglobin >= 8.0 g/dL (may receive red blood cell [RBC] transfusions).
* For patients with solid tumors and known bone marrow metastatic disease:

  * Peripheral absolute neutrophil count (ANC) >= 750/uL
* For patients with solid tumors and known bone marrow metastatic disease:

  * Platelet count >= 50,000/uL
* For patients with solid tumors and known bone marrow metastatic disease:

  * Hemoglobin >= 8.0 g/dL

    * Transfusions are permitted to meet both the platelet and hemoglobin criteria; patients must not be known to be refractory to red blood cell or platelet transfusions
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 or a serum creatinine based on age/gender as follows:

  * 0.6 mg/dL (1 to < 2 years of age)
  * 0.8 mg/dL (2 to < 6 years of age)
  * 1.0 mg/dL (6 to < 10 years of age)
  * 1.2 mg/dL (10 to < 13 years of age)
  * 1.5 mg/dL (male) or 1.4 mg/dL (female) (13 to < 16 years of age)
  * 1.7 mg/dL (male) or 1.4 mg/dL (female) (>= 16 years of age)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) for age
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 110 U/L (for the purpose of this study, the ULN for SGPT is 45 U/L)
* Serum albumin >= 2 g/dL
* Activated partial thromboplastin time (aPTT) =< 1.2 x upper limit of normal

Exclusion Criteria:

* Patients who are pregnant or breast-feeding are not eligible for this study; negative pregnancy tests must be obtained in girls who are post-menarchal; males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method for the duration of study therapy; study drug may also potentially be secreted in milk and therefore breastfeeding women are excluded
* Growth factors that support platelet or white cell number or function must not have been administered within the 7 days prior to enrollment (14 days if pegfilgrastim)
* Patients requiring corticosteroids who have not been on a stable or decreasing dose of corticosteroid for the 7 days prior to enrollment are not eligible
* Patients who are currently receiving another investigational drug are not eligible
* Patients who are currently receiving other anti-cancer agents are not eligible
* Anti-graft-versus-host disease (GVHD) or agents to prevent organ rejection post-transplant:

patients who are receiving cyclosporine, tacrolimus or other agents to prevent either graft-versus-host disease post bone marrow transplant or organ rejection post-transplant are not eligible for this trial

* Patients who have an uncontrolled infection are not eligible
* Patients who have received prior treatment with imetelstat are not eligible
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible
* Patients with prior allogeneic transplants are not eligible

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2014-06-30 (Estimated); Primary Completion 2016-03-25 (Estimated)

PRIMARY OUTCOMES:
Objective response (complete response [CR] or partial response [PR]) according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria or MIBG scoring criteria | Up to 126 days (6 courses)
  Response rates will be calculated as the percent of evaluable patients who are responders, and confidence intervals will be constructed accounting for the two-stage design. Each disease stratum will be reported separately.
Incidence of grade 3 or higher adverse events using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Up to 126 days (6 courses)
  Toxicity tables will be constructed to summarize the observed incidence in each reporting period by type of toxicity and grade. The relative frequency of each type of toxicity will be quantified as the number of toxicity-evaluable cycles in which the adverse event (AE) was noted at grade 3 or higher considered by the treating physician to be possibly, probably or definitely related to one of the agents in the regimen divided by the number of toxicity-evaluable courses administered to patients enrolled on the trial.

SECONDARY OUTCOMES:
Progression-free survival | Date of enrollment until the end progression-free interval (PFI) date, calculated as the date of disease progression, date of death, date of removal of all tumor by surgery or last patient contact, whichever occurs first, assessed up to 3 years
  The probability of remaining progression-free as a function of days since enrollment will be calculated according to the method of Gray accounting for censoring and the competing events.

OTHER OUTCOMES:
Telomerase length by quantitative polymerase chain reaction | Baseline
  The relationship between tumor telomere length and probability of response (as CR or PR) with imetelstat sodium will be assessed using logistic regression.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Thompson, Principal Investigator — Children's Oncology Group